CLINICAL TRIAL: NCT01720355
Title: Pulse Oximetry- Performance During Severe Signal Interference
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0377
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Determine accuracy specifications and labeling claims of a pulse oximeter in a diverse subject population during severe signal interference over a specified saturation range.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18 to 50 years (inclusive).
2. Must undergo a physical examination by a licensed physician, advanced practice nurse or physician assistant, including a 12 lead ECG, a medical history, and a blood test checking complete blood count and screening for sickle cell trait or disease
3. All female volunteers must have a negative urine pregnancy test prior to participation.

Exclusion Criteria:

1. A room-air baseline % modulation < 1.5% on all four fingers on the test hand
2. Pregnancy or lactating women
3. History of syncopal episodes
4. Hypertension (defined as a systolic pressure of >145 mmHg or a diastolic pressure >90 mm Hg on three consecutive readings)
5. Premature ventricular contractions (PVC's) that are symptomatic or occur at a rate of more than 5/minute
6. History of seizures (except childhood febrile seizures) or epilepsy
7. Routine use of tranquilizers and/or excessive anxiety
8. History of frequent headaches or migraines
9. History of stroke
10. Previous injury or trauma to fingers or hands that may change blood flow or vascular supply and affect our ability to test multiple sensors
11. History of "altitude sickness" defined as headaches, malaise or dizziness when in the mountains or in an aircraft at altitude significantly above sea level for a prolonged period of time (> 1 hour)
12. History of significant respiratory disease, such as severe asthma, emphysema, etc.
13. Sickle cell disease or trait.
14. The use of medications, pre-existing medical conditions, treatment for a medical condition or any other reason deemed relevant by the clinician conducting the study.
15. A clinically significant abnormal finding on medical history, physical examination, clinical laboratory test or ECG. Clinical significance will be assessed by the principal investigator or designee.
16. Prior or known allergies to lidocaine (or similar pharmacologic agents, e.g., Novocain)
17. Prior or known allergies to heparin
18. History of transient ischemic attacks or carotid artery disease
19. History of myocardial ischemia, angina, myocardial infarction, congestive heart failure or cardiomyopathy
20. History of chronic renal impairment
21. History of recent arterial cannulation (less than 1 month prior to study)
22. History of complications from previous arterial cannulation
23. Current use of blood thinners

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, well perfused
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
SpO2 Accuracy (percentage of blood oxygen saturation) | 1.5 hours per subject

CONTACTS AND LOCATIONS:
Locations (1):
- Covidien, Boulder, Colorado, United States